CLINICAL TRIAL: NCT03879707
Title: Improving Sleep Quality After Total Joint Arthroplasty ( TJA)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator elected not to proceed with project
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Derek Amanatullah, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49586
Record Dates: First submitted 2019-02-14; First posted 2019-03-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pain After TJA
MeSH Terms: interventions — Melatonin; Magnesium; Tablets

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Melatonin and magnesium for 14 days
  Interventions: Drug: Melatonin 5 mg; Drug: Magnesium 500Mg Oral Tablet
- Control (Placebo Comparator): Placebo for 14 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Melatonin 5 mg — Melatonin is known to induce sleep
  Arms: Experimental
Drug: Placebo Oral Tablet — Placebo
  Arms: Control
Drug: Magnesium 500Mg Oral Tablet — Magnesium plays a role in supporting deep, restorative sleep by maintaining healthy levels of GABA, a neurotransmitter that promotes sleep. Research indicates supplemental magnesium can improve sleep quality, especially in people with poor sleep
  Arms: Experimental

SUMMARY:
The purpose of this study is the evaluate and improve sleep quality after Total joint replacement.

DETAILED DESCRIPTION:
Patients in early stage after TKA tend to suffer from sleep problem. Sleep disturbances frequently occur in patients after surgery, and its occurrence is harmful for postoperative recovery. Many factors can affect the quality of sleep after a major surgery including anesthesia-type, narcotic use and discomfort due to pain or restricted leg movements. Pain directly leads to sleep disruption or even deprivation and, in turn, poor-quality sleep aggravates pain sensation. There seems to be a vicious circle: pain - poor-quality sleep - intensified pain - even poorer-quality sleep.

Presumably, if a patient suffers from catastrophizing, depression and anxiety , the result of TKA will be worse due to poor sleep.

ELIGIBILITY:
Inclusion criteria -Adults 18 years and older

Exclusion criteria -

1. No chronic pain
2. Patients underwent revision or bilateral surgery.
3. Patients underwent fracture.
4. Patients suffering from dementia / delirium
5. Patients on narcotics greater than 10mg hydrocodom before surgery
6. Not willing to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Effect of melatonin and magnesium on pain | 90 days
  Effect of interventions on pain will be measured. It will done at follow up period of 2 wks, 6 wks and 3 months.

SECONDARY OUTCOMES:
Effect of melatonin on daily activities | 90 days
  Effect of interventions daily activities using VAS pain scores. Higher the score. more difficulty in performing daily activities
Effect of melatonin on daily activities | 90 days
  Effect of interventions on daily activities using Hip Disability and Osteoarthritis Outcome ( HOOS ) or Knee Disability and Osteoarthritis Outcome ( KOOS) score. The interval score ranges from 0 to 100 where 0 represents total hip/knee disability and 100 represents perfect hip/knee health
Effect of melatonin on daily activities | 90 days
  Effect of intervention on daily activities using Western Ontario and McMaster Universities Arthritis Index (WOMAC). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Effect of melatonin on daily activities | 90 days
  Effect of intervention on daily activities using Pittsberg sleep quality index. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Effect of melatonin on daily activities | 90 days
  Effect of intervention on daily activities using SF 12 score. The lower the score the more disability

CONTACTS AND LOCATIONS:
Overall Officials: Derek Amanatullah, M.D. PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No